CLINICAL TRIAL: NCT04689841
Title: Influence of Short-term Vojta Therapy on the Gait in Healthy Adult Subjects.
Acronym: V&G
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: NUMEN Foundation (Other)
Collaborators: Universidad Europea de Madrid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Numen2
Record Dates: First submitted 2020-12-28; First posted 2020-12-30 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Gait, Frontal
Keywords: gait; Reflex Locomotion; Core stability; Ontogenesis; Neurorehabilitation; Neurological Disorder
MeSH Terms: conditions — Gait Disorders, Neurologic; Nervous System Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vojta Therapy (Experimental): In Vojta therapy, the therapist selectively presses certain areas of the body, with the patient lying prone, - supine or - lateral. These types of stimuli, in humans of any age, provoke automatically and without their own initiative, that is, without the active voluntary collaboration of the person
  Interventions: Other: Vojta Therapy
- Control Group (Placebo Comparator): In the control group, a placebo intervention is administered, similar to an experimental intervention
  Interventions: Other: placebo

INTERVENTIONS:
Other: Vojta Therapy — Reflex locomotion is activated by the "reflexogenic" pathway. In context with reflex locomotion, the term "reflex" does not represent the mode of neuronal control, but rather refers to defined, "automatic" and always equal motor responses produced by external stimuli, applied therapeutically.
  Other Names: Reflex Locomotion
  Arms: Vojta Therapy
Other: placebo — In the control group, a placebo intervention is administered, similar to an experimental intervention
  Arms: Control Group

SUMMARY:
The patterns of reflex locomotion described by Vojta contain all the basic patterns necessary for gait, which can be observed as partial patterns during normal postural ontogenesis in the first year of life. These patterns are triggered throughout life regardless of age, so they can be activated both in healthy subjects and in the presence of neurological pathology in adult patients.

DETAILED DESCRIPTION:
In reflex locomotion, there is a coordinated and rhythmic activation of the entire skeletal muscles and different circuits of the central nervous system are stimulated. The motor reactions that are triggered regularly and cyclically due to pressure stimuli, from certain starting positions, are completely reproducible and as often as desired, even in the newborn child.

All the movements that appear in the development of the human being in grasping, turning, crawling, standing up and walking, are therefore visibly stimulated. They are, according to Prof. Vojta, present even in children of a developmental stage, in which they do not spontaneously yet possess these capacities.

Through the therapeutic application of reflex locomotion, those muscular functions used unconsciously and necessary for spontaneous daily motor skills are activated in the patient, especially in the spine, but also in the arms and legs, hands and feet and in the face.

ELIGIBILITY:
Inclusion Criteria:

* To be over 18 years old.

Exclusion Criteria:

* Present limitations or permanent or temporary injuries to the locomotor system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2021-09-25 (Estimated); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-05-15 (Estimated)

PRIMARY OUTCOMES:
6 Minutes walk | one month
  walk for 6 minutes measuring the meters walked
EMG surface | two month
  surface electromyography in four muscles

REFERENCES:
- [Derived] Perales-Lopez L, Sanz-Esteban I, Jimenez-Antona C, Serrano JI, San-Martin-Gomez A, Vives-Gelabert X, Cano-de-la-Cuerda R. Automatic gait evoking in healthy adults through Vojta's peripheric somatosensory stimulation: a double-blind randomized controlled trial. J Neuroeng Rehabil. 2024 Oct 1;21(1):174. doi: 10.1186/s12984-024-01470-2. PMID 39354570